CLINICAL TRIAL: NCT03862651
Title: MONET BRIDGE(Maintenance Of aNtiplatElet Therapy in Patients With Coronary Stenting Undergoing Surgery) - (Mantenimento Della Terapia Antiaggregante Nei Pazienti Portatori di Stent Coronarico Candidati a Chirurgia)
Brief Title: Maintenance Of aNtiplatElet Therapy in Patients With Coronary Stenting Undergoing Surgery (MONET BRIDGE)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ospedale Santa Croce-Carle Cuneo (Other)
Responsible Party: Principal Investigator, ROBERTA ROSSINI, Principal Investigator, Ospedale Santa Croce-Carle Cuneo
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MB11-2018
Record Dates: First submitted 2019-02-22; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Platelet Aggregation Inhibitors
Keywords: aNtiplatElet Therapy; cangrelor; randomized; DAPT
MeSH Terms: interventions — cangrelor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cangrelor (Experimental): Cangrelor, 0.75 μg/Kg/min, a cangrelor infusion will be started in addition to SOC when the P2Y12 inhibitor has been discontinued after the need for surgery has been determined. The infusions (cangrelor or matching placebo) will continue throughout the pre-operative period
  Interventions: Drug: Cangrelor
- placebo (No Intervention): patients will receive only standard of care, in which the P2Y12 inhibitor is discontinued after the need for surgery has been determined and a placebo infusion is administered

INTERVENTIONS:
Drug: Cangrelor — Cangrelor is an intravenous analog of adenosine triphospate with a potent, selective and specific affinity for P2Y12 receptors.
  Other Names: KENGREXAL® (cangrelor)
  Arms: Cangrelor

SUMMARY:
The MONET BRIDGE study is designed to assess the use of cangrelor as a platelet-inhibiting bridge for patients who discontinue DAPT before cardiac and non cardiac surgery within 12 months from coronary stent implantation. It seeks to determine if initiation of a prolonged cangrelor infusion maintains effective platelet inhibition after discontinuation of P2Y12 and whether a cangrelor infusion before cardiac and non cardiac procedures is safe.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled study enrolling patients with coronary stent, still on DAPT, undergoing cardiac and non cardiac surgery within 12 months from coronary stent implantation.

The MONET BRIDGE study is designed to assess the use of cangrelor as a platelet-inhibiting bridge for patients who discontinue DAPT before cardiac and non cardiac surgery within 12 months from coronary stent implantation. It seeks to determine if initiation of a prolonged cangrelor infusion maintains effective platelet inhibition after discontinuation of P2Y12 and whether a cangrelor infusion before cardiac and non cardiac procedures is safe.

The primary efficacy objective of this study is to demonstrate that a cangrelor infusion will maintain levels of residual platelet reactivity (PRU < 208) as measured by Accriva VerifyNow® P2Y12 assay.

The main safety objective is to demonstrate that patients receiving cangrelor infusion before cardiac and non cardiac surgery have an acceptable safety profile and can undergo surgery without excessive bleeding peri-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent before initiation of any study related procedures.
2. Be ≥ 18 years of age.
3. Have received any dose of a P2Y12 inhibitor (clopidogrel, ticlopidine, prasugrel, or ticagrelor) at any dose within at least 48 hours prior to randomization.
4. Patients undergoing non deferrable cardiac or non cardiac surgery which requires discontinuation of P2Y12 inhibitor due to a significant bleeding risk.

Exclusion Criteria:

1. Confirmed of suspected pregnancy (if woman of child-bearing potential) or lactating females
2. Active bleeding with evident contraindications to DAPT
3. Patients requiring oral anticoagulant therapy
4. PCI within 1 month
5. Intracranial neoplasm or history of intracranial surgery
6. History of bleeding diathesis
7. Thrombocytopenia (platelet count of less than 100,000/µL)
8. Known International Normalized Ratio (INR) greater than 1.5 at screening.
9. Requirement for dialysis treatment (hemodialysis or peritoneal)
10. Estimated Glomeular filtration rate eGFR <30 ml/min
11. Administration of abciximab within 24 hours of randomization or administration of eptifibitide or tirofiban within 12 hours of randomization
12. Plans to continue oral anticoagulant or P2Y12 inhibitors or cangrelor in the pre-operative period
13. Refusal to receive blood transfusion
14. Receipt of fibrinolytic therapy in the 12 hours preceding randomization
15. Allergy, hypersensitivity, or contraindication to cangrelor, mannitol, sorbitol, or microcrystalline cellulose
16. High likelihood of being unavailable for follow-up
17. Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of randomization
18. Any disease or condition which, in the judgment of the investigator, would place the patient at undue risk by being enrolled in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
LEVEL OF RESIDUAL PLATELET REACTIVITY | 1-2 hours
  Accriva VerifyNow P2Y12 assay

SECONDARY OUTCOMES:
ischemic and hemorrhagic endpoints | 30 days
  Bleeding Academic Research Consortium (BARC) grade > 3

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Moschovitis A, Cook S, Meier B. Percutaneous coronary interventions in Europe in 2006. EuroIntervention. 2010 Jun;6(2):189-94. doi: 10.4244/EIJV7I6A31. PMID 20562067
- [Background] Brilakis ES, Banerjee S, Berger PB. Perioperative management of patients with coronary stents. J Am Coll Cardiol. 2007 Jun 5;49(22):2145-50. doi: 10.1016/j.jacc.2007.02.046. Epub 2007 May 23. PMID 17543633
- [Background] Schouten O, van Domburg RT, Bax JJ, de Jaegere PJ, Dunkelgrun M, Feringa HH, Hoeks SE, Poldermans D. Noncardiac surgery after coronary stenting: early surgery and interruption of antiplatelet therapy are associated with an increase in major adverse cardiac events. J Am Coll Cardiol. 2007 Jan 2;49(1):122-4. doi: 10.1016/j.jacc.2006.10.004. Epub 2006 Dec 18. No abstract available. PMID 17207733
- [Background] Albaladejo P, Marret E, Samama CM, Collet JP, Abhay K, Loutrel O, Charbonneau H, Jaber S, Thoret S, Bosson JL, Piriou V. Non-cardiac surgery in patients with coronary stents: the RECO study. Heart. 2011 Oct;97(19):1566-72. doi: 10.1136/hrt.2011.224519. Epub 2011 Jul 26. PMID 21791513
- [Background] Rossini R, Musumeci G, Capodanno D, Lettieri C, Limbruno U, Tarantini G, Russo N, Calabria P, Romano M, Inashvili A, Sirbu V, Guagliumi G, Valsecchi O, Senni M, Gavazzi A, Angiolillo DJ. Perioperative management of oral antiplatelet therapy and clinical outcomes in coronary stent patients undergoing surgery. Results of a multicentre registry. Thromb Haemost. 2015 Feb;113(2):272-82. doi: 10.1160/TH14-05-0436. Epub 2014 Oct 2. PMID 25274620